CLINICAL TRIAL: NCT02089126
Title: A Multicenter, Randomized, Placebo-controlled, Parallel Group, Double-blind, Phase III Trial to Evaluate the Efficacy and Safety of Gemigliptin 50mg qd Added to Ongoing Glimepiride as Fix-dose Combination in Patients With Type 2 Diabetes Inadequately Controlled on Glimepiride Alone
Brief Title: Phase III Trial to Evaluate the Efficacy and Safety of Gemigliptin 50mg qd Added to Ongoing Glimepiride as Fix-dose Combination in Patients With Type 2 Diabetes
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: LG Life Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: LG-GGCL001
Record Dates: First submitted 2014-03-13; First posted 2014-03-17 (Estimated); Last update posted 2014-03-17 (Estimated); Status verified 2014-03

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — LC15-0444

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Gemigliptin/Glimepiride combination (Experimental): Gemigliptin 50mg qd added to ongoing Glimepiride as fix-dose combination. The subjects will take a total of 2 tablets, Gemigliptin/Glimepiride combination & Placebo for Glimepiride.
  Interventions: Drug: Gemigliptin/Glimepiride combination
- Placebo (Placebo Comparator): The subjects will take a total of 2 tablets, Placebo for Gemigliptin/Glimepiride combination & Glimepiride.

INTERVENTIONS:
Drug: Gemigliptin/Glimepiride combination
  Arms: Gemigliptin/Glimepiride combination

SUMMARY:
The study objective is to demonstrate the superiority and safety of the combination therapy (as a fix-dose combination) with Gemigliptin and Glimepiride, compared to the Glimepiride monotherapy in patients with type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with type 2 diabetes
2. Adults who are at least 19 years old
3. Patients who have taken Glimepiride at a stable dose (≥4mg/day) for 8 weeks or more before Visit 1 (screening) as monotherapy or Patients who have taken Glimepiride at a stable dose (≥4mg/day) and Metformin for 8 weeks or more before Visit 1 (screening) as combination therapy
4. Patients who satisfy the following HbA1c (%) criteria: 7 ≤ HbA1c ≤ 11
5. Patients who have been provided an explanation about the objective, method, effects, etc. of the clinical trial and whose informed consent form has been signed by himself/herself or his/her representative
6. Patients who fall under one of the following 3 cases

   1. Patients who are surgically sterile
   2. Post-menopausal females who are above 45 years of age and 2 years after the last menstruation
   3. Fertile premenopausal female patients or male patients without having a surgical sterilization, who have agreed to use at least two contraception methods (one of the barrier methods must be included) for up to 14 days after the administration of the last investigational product to avoid pregnancy.

Exclusion Criteria:

1. Patients with type 1 diabetes, diabetic ketoacidosis, diabetic coma and pre-coma
2. Patients with gestational diabetes or secondary diabetes
3. Patients with NYHA Class III, IV congestive heart failure or arrhythmias requiring treatment
4. Patients with thyroid gland dysfunction and TSH that is out of normal range
5. Patients with pituitary insufficiency or adrenal insufficiency
6. Patients with hereditary problems, such as galactose intolerance, Lapp lactose deficiency or glucose-galactose malabsorption
7. Female patients who are pregnant or breastfeeding
8. Patients whose BMI exceeds 40 kg/m2
9. Patients whose creatinine clearance is below 30mL/min/1.73m2
10. Patients whose bilirubin level exceeds 1.5 times the upper limit of the normal range and whose ALT/AST level exceeds 2.5 times the upper limit of the normal range
11. Patients who are continuously taking the following drugs for 2 weeks or more at Visit 1 (screening), or need to take them continuously and repeatedly

    * cyclosporin, sirolimus, tacrolimus, nicotinic acid (≥1500mg/day), isotretinoin
    * Strong CYP3A4 inducers: rifampicin (rifampin), phenytoin, carbamazepine, rifabutin, phenobarbital
    * warfarin, dicoumarin, digoxin
    * systemic glucocorticoids
12. Patients who have taken anti-obesity drugs or had a surgery related to obesity within 12 weeks before Visit 1 (screening)
13. Patients who have received insulin and GLP-1 analogue treatment within 8 weeks prior to Visit 1 (screening)
14. Patients who have received a treatment due to malignant tumor within 5years before Visit 1 (screening) However, patients whose basal cell or squamous cell skin cancer or in situ cervical cancer has been treated can be enrolled.
15. Patients with a history of myocardial infarction, unstable angina and coronary artery bypass surgery within 6 months prior to Visit 1 (screening)
16. Patients with a history of alcohol or drug addiction within 1 year prior to Visit 1 (screening)
17. Patients who have a medical history of hypersensitivity to the same class as Gemigliptin or dipeptidyl peptidase 4 (DPP 4) inhibitor drugs
18. Patients with a history of hypersensitivity to the drugs belonging to the same class as Glimepiride or sulfonylureas and sulfonamide
19. Patients who have participated in another clinical trial within 3 months prior to Visit 1 (screening)
20. Patients deemed unsuitable for this trial based on the judgment of the investigator

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 230 (Estimated)
Dates: Start 2014-06; Primary Completion 2016-09 (Estimated)

PRIMARY OUTCOMES:
HbA1c Changes | Week 0, Week 24

CONTACTS AND LOCATIONS:
Locations (1):
- The Catholic University of Korea Seoul St. Mary's Hospital, Seoul, South Korea